CLINICAL TRIAL: NCT04326387
Title: Evaluation of Novel Diagnostic Tests for 2019-nCOV
Brief Title: Evaluation of Novel Diagnostic Tests for COVID-19
Acronym: COVIDx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Prof. Ravindra Gupta, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: COVIDx
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Acute Disease; Coronavirus; Respiratory Viral Infection
Keywords: Coronavirus; COVID-19; nCOV-2019
MeSH Terms: conditions — Acute Disease; Coronavirus Infections; COVID-19 | interventions — Diagnosis; Diagnostic Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Throat/Nasal Swab, Nasopharyngeal Swab, Endotracheal tube aspirate and whole blood-serum for viral-RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research Participants (Patients): Inpatients symptomatic of suspected COVID-19 Baseline swab of nose/throat, nasopharyx, or endotracheal tube aspirate. SAMBA II point of care test on this swab.
  Standard of care bloods taken for PHE and additional confirmatory diagnostic PCR assessment.
  Serum antibody tests on any excess blood tests during inpatient stay for immune response monitoring.
  Outcome assessment at 1 month
  Interventions: Diagnostic Test: SAMBA II (Diagnostic for the Real World); Diagnostic Test: Public Health England Gold Standard; Diagnostic Test: Cambridge Validated Viral Detection Method; Diagnostic Test: Radiological Detection

INTERVENTIONS:
Diagnostic Test: SAMBA II (Diagnostic for the Real World) — Point of care Isothermal-PCR Viral RNA Amplication for virus detection
Diagnostic Test: Public Health England Gold Standard — Reverse Transcription PCR
Diagnostic Test: Cambridge Validated Viral Detection Method — Reverse Transcription PCR
Diagnostic Test: Radiological Detection — Chest X-ray & CT Scan detection of viral infection in the lungs
  Other Names: Chest X-ray, CT Scan

SUMMARY:
COVID-19 (also known as Coronavirus) originated in the Wuhan China and has since spread to at least 159 countries around the world. It was declared a pandemic by the World health organisation on the 11th of March 2020. The cases in the United Kingdom continue to increase exponentially with up to 5 683 people diagnosed as on the 22nd of March 2020. It is estimated that 1 in 5 people diagnosed will require hospital admission and 1 in 20 intensive care treatment. By developing and improving diagnostic testing, we can accurately diagnose infected cases to triage appropriate treatments, identify individuals for quarantine in order to prevent transmission and obtain information regarding patient's immune systems.

At present, the diagnostic test is a highly specific method of genetic amplification called 'Reverse Transcription - Polymerase Chain Reaction' or RT-PCR, which allows detection of very small amounts of genetic mutations caused by the COVID-19 virus. However, this method must be completed in highly specialised facilities, which are few and far between, increasing time to diagnosis (currently 48-72 hours), increasing exposure to non-infected individuals, and overburdening the analysing facilities. The ideal solution is a point of care (POC) test that can give results immediately. This study aims to harness the point of care technology of the SAMBA II device (Diagnostics for the Real World Ltd.), which is a CE-marked device that has been used with success in the identification of Human Immunodeficiency Virus (HIV), by amplifying genetic material without the need to increase and decrease temperatures during the amplification process.

In the COVIDx study, 200 patients meeting the Public Health England's (PHE) inpatient definition of having suspected COVID-19 will be approached, consented and a sample from throat and nasal swab (combined) or tracheal fluid taken and tested using the SAMBA II method. A combination of the standard PHE RT-PCR and an additional validated laboratory PCR technique will be used as a control in line with standard clinical practice. Patients will undergo an additional serum tests on existing samples as made available after routine clinical assessments to monitor antibody response. Patients will be followed for clinical outcomes at 28 days post-admission.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or above
* Patient requiring hospital admission AND AT LEAST ONE OF
* Clinical or Radiological evidence of pneumonia
* Acute respiratory distress syndrome
* Influenza like illness (defined as fever >37.8oC and at least one of the following respiratory symptoms, which much be of acute onset: persistent cough (with or without sputum), hoarseness, nasal discharge or congestion, shortness of breath, sore throat, wheezing, sneezing)

Exclusion Criteria:

* Patients who have not had the standard PHE COVID-19 test applied
* Unwilling or unable to comply with research swab of nose & throat or tracheal fluid

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who meet current PHE hospital inpatient definition of possible case of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-04-07 (Estimated); Study Completion 2021-10-07 (Estimated)

PRIMARY OUTCOMES:
SAMBA COVID-19 POC PCR Test | 28 days
  Measuring the diagnostic accuracy of the SAMBA II POC-sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) tested against a dual composite reference standard

SECONDARY OUTCOMES:
Patient acceptability | 28 days
  Evaluating the participant acceptability of the SAMBA swab intervention using a participant reported discomfort scale
Immune Response Positivity | 40 days
  Time to positive IgM/IgG test positivity

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra Prof. Gupta, BMBCh, Principal Investigator — University of Cambridge & Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided